CLINICAL TRIAL: NCT06887803
Title: A Phase I/II Open-Label, Multi-centre Study to Assess the Safety and Tolerability of Roginolisib in Combination With Ruxolitinib in Patients With Myelofibrosis (MF) Who Are Unresponsive to an Approved JAK Inhibitors (HEMA-MED)
Brief Title: A Study of Roginolisib in Combination With Ruxolitinib in Patients With Myelofibrosis (MF) Who Are Unresponsive to JAK Inhibitors
Acronym: HEMA-MED
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: iOnctura (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOA-244-203; 2024-515252-20 (EudraCT Number)
Record Dates: First submitted 2025-02-26; First posted 2025-03-20 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Myelofibrosis (MF)
Keywords: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Intervention Model Description: Single Arm, open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Roginolisib and ruxolitinib
  Interventions: Drug: Roginolisib

INTERVENTIONS:
Drug: Roginolisib — IOA-244: 80 mg (corresponding to 72 mg roginolisib) Ruxolitinib: up to 25 mg BD

SUMMARY:
The goal of this clinical trial is to learn how roginolisib works in comparison to standard treatment in adult patients with Myelofibrosis. The main questions it aims to answer is to evaluate the safety and tolerability of roginolisib when administered in combination with ruxolitinib.

DETAILED DESCRIPTION:
A Phase I/II Open-Label, Single Arm Multi-centre Study to Assess the Safety and Tolerability of Roginolisib in Combination with Ruxolitinib in Patients with Myelofibrosis (MF) who are Unresponsive to JAK inhibitors (HEMA-MED).

This study will enrol approximately 26 male and female patients aged over 18 years with MF, who have been treated with ruxolitinib for ≥ 3 months with a stable dose ≥ 10 mg for at least the last 8 weeks prior to Day 1 and no significant spleen reduction.

The study will initially enrol 13 patients in Part 1 to assess the benefit/risk profile of roginolisib when combined with ruxolitinib. Part 2 will enrol an additional 13 patients to further characterize the benefit/risk.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age inclusive, at the time of signing the informed consent.
2. Capable of giving signed informed consent, which includes compliance with the requirements of this protocol.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
4. Diagnosis of MF, Post-Polycythaemia Vera Myelofibrosis MF (PPV-MF), or post-essential thrombocythemia MF (PET-MF)
5. Dynamic International Prognostic Scoring System (DIPSS) risk category of intermediate-1, intermediate-2, or high
6. Treated with ruxolitinib for ≥ 3 months with a stable dose ≥ 10 mg for a minimum of 8 weeks prior to Day 1. Furthermore, patients must show an unsatisfactory spleen reduction, such as a reduction of less than 25%, and spleen must be palpable ≥ 10 cm below the left costal margin on physical examination
7. Did not receive experimental drug therapy for MF or any other drug considered as an effective treatment for MF (e.g., danazol, hydroxyurea, interferon products) with the exception of ruxolitinib, within 3 months of starting study drug (except in conditions where other effective treatments for MF were completed 6 months prior to starting ruxolitinib)
8. Independent of spleen size, active symptoms of MF at the screening visit, as demonstrated by the presence of a Total Symptom Score (TSS) of ≥ 10 using the Screening Symptom Form.
9. Peripheral blast count < 10%
10. Act to avoid pregnancy or fathering children based on the criteria below:

    1. Women of non-childbearing potential (i.e., surgically sterile with a hysterectomy and/or bilateral oophorectomy OR ≥ 12 months of amenorrhea and at least 50 years of age).
    2. Women of childbearing potential who had a negative serum pregnancy test at screening and who agree to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through safety follow-up, at least 1 month after the last dose of study treatment. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the patient and their understanding confirmed.
    3. Men who agree to take appropriate precautions to avoid fathering from screening through safety follow-up, at least 1 month after the last dose of study treatment. Permitted methods that are at least 99% effective in preventing pregnancy (see Appendix 3) should be communicated to the patient and their understanding confirmed.

Exclusion Criteria:

1. Inability to swallow food or any condition of the upper gastrointestinal tract that precludes administration of oral medications.
2. History of a prior Grade 3 or 4 AE which did not respond to therapy or resolved with treatment interruptions and returned to at least Grade 1, other than fatigue. Note: Patients with ≤ Grade 2 neuropathy or alopecia are an exception and may enrol.
3. Active autoimmune process (e.g., rheumatoid arthritis, moderate or severe psoriasis, multiple sclerosis, inflammatory bowel disease, immune colitis) for which systemic treatment (i.e., use of disease-modifying agents, corticosteroids, or immunosuppressive drugs) is required. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
4. History or presence of an abnormal ECG that, in the Investigator's opinion, is clinically meaningful. Screening QTc interval > 480 milliseconds is excluded (corrected by Fridericia). In the event that a single QTc is > 480 milliseconds, the patient may enrol if the average QTc for the 3 ECGs is < 480 milliseconds. For patients with an intraventricular conduction delay (QRS interval > 120 msec), the JTc interval may be used in place of the QTc with Sponsor approval. The JTc must be < 340 milliseconds if JTc is used in place of the QTc. Patients with left bundle branch block are excluded.
5. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrolment), myocardial infarction (< 6 months prior to enrolment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
6. Patients with active malignancy requiring concurrent intervention or previous malignancies unless a complete remission was achieved at least 2 years prior to study entry and no additional therapy is required during the study period and the patient is assessed at low risk of relapse by the investigator. Note: Patients with a slow progressing cancer (e.g. prostate) or an in situ cancers (e.g. cervical dysplasia) are permitted.
7. Any serious or uncontrolled medical disorder or active infection that, in the opinion of the Investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the patient to receive protocol therapy.
8. Use of the following treatments within the time periods noted:

   1. Erythropoiesis stimulating agent (ESA) within 4 weeks prior to start of roginolisib.
   2. Splenic irradiation within 3 months prior to start of roginolisib.
9. Major surgery within 2 weeks of the first dose of study drug (minimally invasive procedures such as bronchoscopy, bone marrow biopsy, insertion of a central venous access device, and insertion of a feeding tube are not considered major surgery and are not exclusionary)
10. Receiving an immune-suppressive based treatment for any reason (including chronic use of systemic corticosteroid at doses > 10 mg/day prednisone equivalent) within 14 days prior to the first dose of study treatment. Use of inhaled or topical steroids (including but not limited to creams or intra-articular injection) or brief corticosteroid use for radiographic procedures or systemic corticosteroids ≤ 10 mg is permitted.
11. Have received a live vaccine within 30 days of planned start of study therapy while on trial. Other type of vaccines, including SARS-Co2 vaccines, are allowed.
12. Known allergy or reaction to any component of either study drugs or formulation components.
13. Currently breastfeeding.
14. Known alcohol or other substance abuse.
15. Laboratory and medical history parameters not within Protocol-defined range.

    1. Absolute neutrophil count < 1.5 × 109/L.
    2. Platelet count < 100 × 109/L.
    3. Haemoglobin < 8 g/dL (transfusion is acceptable to meet this criterion).
    4. Serum creatinine ≥ 1.5 × institutional ULN or measured or calculated creatinine clearance (glomerular filtration rate can also be used in place of creatinine or CrCl) < 50 mL/min for patients with creatinine levels > 1.5 × institutional ULN.
    5. Aspartate aminotransferase (AST) or Alanine transaminase (ALT) ≥ 2.5 × ULN in the absence of hepatic metastases or ≥ 5 × ULN with hepatic metastases at screening.
    6. Total bilirubin ≥ 1.2 × ULN are excluded unless direct bilirubin is ≤ ULN. If there is no institutional ULN, then direct bilirubin must be < 40% of total bilirubin to be eligible (except patients with Gilbert syndrome, who must have total bilirubin < 51.3 μmol/L).
    7. International normalized ratio or prothrombin time (PT) > 1.5 × ULN.
    8. Activated partial thromboplastin time (aPTT) > 1.5 × ULN.
    9. Evidence of acute infection of hepatitis B virus (HBV), (for example: positive for HBsAg, anti-HBc, IgM anti-HBc and negative for anti-HBs), hepatitis C virus (HCV) (for example: HCV antibody reactive; HCV RNA detected) and HIV.

    Patients who are on stable antiviral therapy, in good clinical control (ie for HIV a viral load < 400 copies/mL and a CD4+ count of ≥ 350 cells/uL) AND asymptomatic are eligible for the study
16. Presence of active or inactive 'latent' tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events | Day 1 and 15 of cycle 1; Day 1 of each subsequent cycle whilst on treatment anticipated to be 52 weeks. Cycle length 28 days
  Safety measure by Adverse Event's
Number of Participants with abnormal ECG recordings | Day 1 of each cycle whilst on treatment anticipated to be 52 weeks. Cycle length 28 days
  Changes observed on 12-lead ECG
Number of participants with abnormal laboratory parameters | Day 1 and 15 of cycle 1; Day 1 of each subsequent cycle whilst on treatment anticipated to be 52 weeks. Cycle length 28 days
  Standard laboratory parameters (including clinical chemistry, heamatology)
Number of participants with changes in blood pressure measurements | Day 1 and 15 of cycle 1; Day 1 of each subsequent cycle whilst on treatment anticipated to be 52 weeks. Cycle length 28 days
  As measured by blood pressure measurements

SECONDARY OUTCOMES:
To evaluate biomarker responses (e.g., Treg reduction) when roginolisib is administered in combination with ruxolitinib in patients with MF. | Day 1 of Cycle 1, 2 and 3 and then Day 1 of every other cycle (C5, C7 etc) until end of treatment anticipated to be 52 weeks. Cycle length is 28 days
  Changes in peripheral blood Tregs from baseline at Week 12 and continued reduction over time
Spleen reduction responses of roginolisib when administered in combination with ruxolitinib in patients with MF. | Splenic response rate at baseline, 12 and 24 weeks. Duration of spleen response every 12 weeks whilst on treatment anticipated to be 52 weeks.
  Splenic response rate (SRR) of ≥15%, ≥25% and ≥35% reduction in spleen volume as assessed by MRI/CT
  Duration of spleen response
To evaluate preliminary signs of clinical efficacy of roginolisib when given in combination with ruxolitinib | Patients will be followed up for overall survival every 12 weeks, for 96 weeks from last patient enrolled, until their death or end of the study
  Proportion of patients with transfusion independence at 12 and 24 weeks where applicable
To determine the improvements of MF related symptoms when roginolisib is given in combination with ruxolitinib as assessed by the Myelofibrosis Symptom Assessment Form (MFSAF) | TTS and MFSAF measured at baseline and at 12 and 24 weeks.
  Proportion of patients who have any reduction in Total Symptom Score (TSS) at 12 and 24 weeks compared to baseline as measured by Myelofibrosis Symptom Assessment Form (MFSAF) Proportion of patients who have a reduction of ≥25% and ≥50% in TSS as measured by Myelofibrosis Symptom Assessment Form (MFSAF) Mean change in TSS as measured by Myelofibrosis Symptom Assessment Form (MFSAF) Time to the first ≥50% reduction compared to baseline in TSS as measured by Myelofibrosis Symptom Assessment Form (MFSAF) Duration of TSS response as measured by MFSAF (e.g., duration of TSS ≥25% and ≥50%)
To determine the pharmacokinetic (PK) parameters of roginolisib when given in combination with ruxolitinib to allow exposure/response and/or exposure/safety assessment | Day 1 of each cycle whilst on treatment anticipated to be 52 weeks. Cycle length 28 days
  Concentration of roginolisib at pre-dose and steady state levels Area under the curve [AUC]
To evaluate preliminary signs of clinical efficacy of roginolisib when given in combination with ruxolitinib | Patients will be followed up for overall survival every 12 weeks, for 96 weeks from last patient enrolled, until their death or end of the study
  Overall Survival (OS) defined as the time from the date of the first dose of study treatment until death from any cause anticipated

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lahn, Dr, Study Director — iOnctura
Locations (7):
- Italy (4):
  - Azienda Ospedaliero Universitaria Careggi Firenze, Struttura Complessa di Ematologia, Florence, Florence
  - IRCCS Clinical Institute Humanitas, Rozzano, Milan
  - Istituto di Ematolgia e Oncologia Medica, Bologna
  - Azienda Sanitario Universitaria Friuli Centrale, Udine
- Spain (3):
  - Vall d'Hebron University Hospital, Barcelona
  - Avigunda Gran via de l'Hospitalet 199-203, 08908 L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: Undecided